CLINICAL TRIAL: NCT02478853
Title: Agir Sur Sa SantE- Impact of a Regional Integrated Prevention and Management of Cardio-metabolic Chronic Diseases Program in Primary Care
Brief Title: Impact of a Regional Program Agir Sur Sa SantE
Status: Active, not recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: CCER 14-15 -15
Record Dates: First submitted 2015-04-20; First posted 2015-06-23 (Estimated); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus, Type 2; Obesity; Hypertension; Dyslipidemias; Cardiovascular Diseases; Smoking
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Hypertension; Dyslipidemias; Cardiovascular Diseases; Smoking

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Implementation of a new regional care framework — Integrated care framework for the prevention and management of cardio-metabolic chronic diseases in primary care

SUMMARY:
The prevention and control of lifestyle-related non-communicable chronic diseases, including diabetes, obesity and cardiovascular disorders, that share common risk factors, has now become a major focus of the World Health Organization. Lifestyle modification, like improvement of diet, physical activity and tobacco cessation, is the corner stone of diabetes and cardio-metabolic chronic diseases (CMCD) prevention and management. Under the leadership of decision-makers of our regional health Agency in order to improve accessibility and quality of care, our team has collaborated to the development and implementation of an integrated care framework for the prevention and management of cardio-metabolic chronic diseases in primary care. This new care framework is currently being implemented in the context of community health centers (fall 2014) and family medicine groups (spring 2015), with the support of a Quebec Ministry of Health grant. The current research proposal aims to evaluate the implementation of this new care framework and explore its impact in the primary care context. This project is very important as it will generate knowledge on new models of care integrating preventive and management interventions in primary care settings, in continuum with specialized health care services and their implementation in an entire region.

DETAILED DESCRIPTION:
BACKGROUND: In an era where cardio-metabolic chronic diseases (CMCD) take epidemic proportions, health systems have to react by providing care to manage but also to prevent them. Our region has demonstrated leadership in developing and implementing regional care frameworks and patient trajectories defining services throughout the continuum of care (from community to primary to specialized care). However, these diabetes, cardiac rehabilitation and 0-5-30 prevention programs have been implemented in silos. Under the leadership of decision-makers of our regional health Agency, in order to improve accessibility and quality of care, our team has worked on the development and implementation of an integrated care framework for the prevention and management of cardio-metabolic chronic diseases: Agir Sur Sa SantÉ (ASSSÉ). This new framework, based on individual/group motivational techniques, care protocols and collective orders, is currently being implemented in the context of community health centers (CSSS). The investigators recently received a Quebec Ministry of Health grant to continue supporting the implementation in CSSS, implement the care framework in family medicine groups (FMG; spring 2015) and initiate some baseline evaluations (satisfaction and perceptions questionnaires). The investigators hypothesize that successful implementation of ASSSÉ could improve accessibility indicators, for patients affected or at risk for CMCD, patient and primary care personnel satisfaction, fidelity, quality and continuity of care in the context of FMGs.

OBJECTIVES: The investigators aim to:

1. Analyze the implementation process of the new ASSSÉ framework in the context of FMGs by: a) establishing its acceptability and perceived usefulness by patients and health professionals; b) identifying the determinants (barriers and facilitators) of its implementation; c) describing the strategies used to implement the ASSSÉ care framework in FMGs.
2. Estimate the size of the effects of ASSSÉ (including main effects and variability of effects across FMGs to allow for informed sample size calculation in the planning of a future large-scale trial) on: a) patients (satisfaction, health outcomes); b) primary care professionals (practice, satisfaction, self-efficacy); c) health care system (organizational and technical quality of care indicators, accessibility and continuity of care indicators, fidelity of care to framework).
3. Effectively share knowledge obtained through these activities to relevant stakeholders in the health care and public health sectors, including policy makers, decision makers, health care professionals and patients using innovative tools and approaches.

METHODS AND APPROACH: This participatory research project will use a mixed-method approach combining qualitative and quantitative assessments. The project will be conducted in three steps: 1-Pre-implementation evaluation: Services and patient trajectories currently provided in all 14 FMGs of the Eastern Townships will be assessed using chart reviews to evaluate technical quality of care indicators and health outcomes. The investigators will also use questionnaires evaluating the concordance with the Expended chronic care model, self-efficacy, satisfaction of personnel and patients, and potential areas to target for improvement to assess organizational quality of care. Questionnaires and semi-structured group interviews with health professionals, decision-makers and patients with, or at risk for, CMCD will also be performed; 2- Post-implementation evaluation and data analysis: 12, 24 and 36 months after initiation of implementation, the investigators will perform a similar evaluation as done in the initial phase. Semi-structured group interviews will only be repeated at 24 months. Pre- and post-implementation comparisons will be performed using paired t-tests for continuous variables and McNemar tests for dichotomous variables to identify areas of improvement and persistent gaps. 3-Knowledge translation(KT): Integrated KT is an important outcome of this research, has already begun and will occur throughout the project with the various actors involved. The investigators will also reach out to various target audiences (health professionals, decision-makers and policy-makers, patients and Canadian population) through classic end-of-grant KT and the production of a clear executive summary of research results.

IMPACT: Considering the epidemic of chronic diseases, this project is very important as it will generate knowledge on models of care integrating preventive and management interventions of multiple conditions in primary care, in continuum with specialized health care services. It also has high transferability potential in various provincial and disease contexts.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals involved in CMCD management in the targeted clinics
* Eligible patients should have at least one CMCD (diabetes, pre-diabetes, obesity, cardio- or cerebrovascular disease, hypertension, dyslipidemia) or be active smokers.

Exclusion Criteria:

* Patients who are not able to fill out questionnaires with help

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All healthcare professionals involved in CMCD management in the targeted clinics will be invited to participate (questionnaires and group interviews). All adult patients prospectively presenting at the targeted clinics will receive an invitation letter describing the project.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-12 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Implementation of the new care framework assessed with interviews, chart audit and questionnaires | 36 months
  Investigators will assess implementation of the framework including barriers and facilitators, acceptability and perceived usefulness and the strategies used to implement

SECONDARY OUTCOMES:
Patients' satisfaction measure with questionnaire | 36 months
  Patients' satisfaction
Patients' health outcome measure with chart audit | 36 months
  Health outcome such as weight, HbA1c,...
Primary care professionals' satisfaction measure with questionnaire | 36 months
  Primary care professionals' satisfaction
Primary care professionals' practice measure with interviews | 36 months
  Primary care professionals' practice
Primary care professionals' self-efficacy measure with questionnaire | 36 months
  Primary care professionals' self-efficacy
Organizational quality of care indicators measure with questionnaire | 36 months
  Organizational quality of care indicators
Technical quality of care indicators measure with chart audit | 36 months
  Technical quality of care indicators
Accessibility of care indicators measure with administrative data | 36 months
  Accessibility of care indicators
Continuity of care indicators measure with chart audit | 36 months
  Continuity of care indicators
Fidelity of care to framework measure with chart audit | 36 months
  Fidelity of care to framework

CONTACTS AND LOCATIONS:
Overall Officials: Marie-France Langlois, MD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du CHUS, Sherbrooke, Quebec, Canada